CLINICAL TRIAL: NCT04815148
Title: A Phase Ia/Ib Study to Evaluate the Safety, Tolerability and PK of MH004 Topical Cream in Healthy Adult Volunteers and to Investigate Its Efficacy and Safety Profile in Participants With Atopic Dermatitis or Rheumatoid Arthritis
Brief Title: MH004 Topical Cream in Healthy Adult Volunteers and Participants With Atopic Dermatitis or Rheumatoid Arthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minghui Pharmaceutical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MH004-CP001EN
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Atopic Dermatitis; Rheumatoid Arthritis
MeSH Terms: conditions — Dermatitis, Atopic; Arthritis, Rheumatoid

STUDY DESIGN:
Masking Description: Phase Ia is open label while Phase Ib is double blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Phase Ia: MH004 (0.1%) in healthy volunteers (Experimental): SAD and MAD
  Interventions: Drug: MH004 Ia(0.1%)
- Phase Ia: MH004 (0.3%) in healthy volunteers (Experimental): SAD and MAD
  Interventions: Drug: MH004 Ia(0.3%)
- Phase Ia: MH004 (1%) in healthy volunteers (Experimental): SAD and MAD
  Interventions: Drug: MH004 Ia(1%)
- Phase Ia: MH004 (3%) in healthy volunteers (Experimental): SAD and MAD
  Interventions: Drug: MH004 Ia(3%)
- Phase Ib-1: MH004 (0.1%) in Atopic Dermatitis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Atopic Dermatitis
  Interventions: Drug: MH004 Ib-1(0.1%)
- Phase Ib-1: MH004 (0.3%) in Atopic Dermatitis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Atopic Dermatitis
  Interventions: Drug: MH004 Ib-1(0.3%)
- Phase Ib-1: MH004 (1%) in Atopic Dermatitis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Atopic Dermatitis
  Interventions: Drug: MH004 Ib-1(1%)
- Phase Ib-2: MH004 (0.3%) in Rheumatoid Arthritis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Rheumatoid Arthritis
  Interventions: Drug: MH004 Ib-2(0.3%)
- Phase Ib-2: MH004 (1%) in Rheumatoid Arthritis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Rheumatoid Arthritis
  Interventions: Drug: MH004 Ib-2(1%)
- Phase Ib-2: MH004 (3%) in Rheumatoid Arthritis (Experimental): 28-Day Repeated Dosing in Participants with Mild to Moderate Rheumatoid Arthritis
  Interventions: Drug: MH004 Ib-2(3%)

INTERVENTIONS:
Drug: MH004 Ia(0.1%) — Spread approx. 1 g of MH004 topical cream to the upper thigh skin.
  Other Names: MH004 Topical Cream
  Arms: Phase Ia: MH004 (0.1%) in healthy volunteers
Drug: MH004 Ia(0.3%) — Spread approx. 1 g of MH004 topical cream to the upper thigh skin.
  Other Names: MH004 Topical Cream
  Arms: Phase Ia: MH004 (0.3%) in healthy volunteers
Drug: MH004 Ia(1%) — Spread approx. 1 g of MH004 topical cream to the upper thigh skin.
  Other Names: MH004 Topical Cream
  Arms: Phase Ia: MH004 (1%) in healthy volunteers
Drug: MH004 Ia(3%) — Spread approx. 1 g of MH004 topical cream to the upper thigh skin.
  Other Names: MH004 Topical Cream
  Arms: Phase Ia: MH004 (3%) in healthy volunteers
Drug: MH004 Ib-1(0.1%) — Spread approx. 0.5 g of MH004 topical cream to the area of Target AD Lesions.
  Other Names: MH004 Topical Cream
  Arms: Phase Ib-1: MH004 (0.1%) in Atopic Dermatitis
Drug: MH004 Ib-1(0.3%) — Spread approx. 0.5 g of MH004 topical cream to the area of Target AD Lesions.
  Other Names: MH004 Topical Cream
  Arms: Phase Ib-1: MH004 (0.3%) in Atopic Dermatitis
Drug: MH004 Ib-1(1%) — Spread approx. 0.5 g of MH004 topical cream to the area of Target AD Lesions.
  Other Names: MH004 Topical Cream
  Arms: Phase Ib-1: MH004 (1%) in Atopic Dermatitis
Drug: MH004 Ib-2(0.3%) — Spread approx. 0.5 g of MH004 topical cream to the Target Joint.
  Other Names: MH004 Topical Cream
  Arms: Phase Ib-2: MH004 (0.3%) in Rheumatoid Arthritis
Drug: MH004 Ib-2(1%) — Spread approx. 0.5 g of MH004 topical cream to the Target Joint.
  Other Names: MH004 Topical Cream
  Arms: Phase Ib-2: MH004 (1%) in Rheumatoid Arthritis
Drug: MH004 Ib-2(3%) — Spread approx. 0.5 g of MH004 topical cream to the Target Joint.
  Other Names: MH004 Topical Cream
  Arms: Phase Ib-2: MH004 (3%) in Rheumatoid Arthritis

SUMMARY:
This is a Phase Ia/Ib Study of MH004 in Healthy Adult Volunteers, participants with Mild to Moderate Atopic Dermatitis and participants with Mild to Moderate Rheumatoid Arthritis.

DETAILED DESCRIPTION:
The study includes 2 parts:The first part (Phase Ia) is a single ascending dose (SAD) study and a multiple ascending dose (MAD) study in healthy volunteers. The second part (Phase Ib) includes two randomised, Placebo-Controlled 28-day repeated dose studies for AD and RA participants respectively, using defined concentrations of the topical cream based on the PK and safety data in healthy volunteers in Phase Ia.

ELIGIBILITY:
Inclusion Criteria:

Phase Ia and Ib:

1. Phase Ia: Adults, age 18 - 45 years old, inclusive, at time of screening. Phase Ib: Adults, age 18 - 70 years old, inclusive, at time of screening.
2. Willing and able to understand and sign an informed consent form and to comply with all aspects of the protocol.
3. Participants whose body mass index (BMI) at screening is within a range of ≥ 18.5 kg/m2 and <35 kg/m2.

   (BMI = Body Weight (kg) / [Height (m) × Height (m)])
4. Has abstained from smoking or use of tobacco products from 6 months prior to study drug administration and for the entire duration of the study.
5. Participant's medical history shows no contraindication to JAK inhibitors.
6. Participants judged to be in good health by the Investigator based upon the results of physical examinations (PEs), 12-lead electrocardiogram (ECG) test, and all items of routine laboratory tests, including serum biochemistry, hematology and urinalysis, are within normal range, or if outside normal range they are deemed not clinically significant as judged by the Investigator. Assessment items of blood biochemistry include albumin, total protein, total bilirubin, ALP, SGOT, SGPT, BUN, serum creatinine, CK and fasting lipid profile (total cholesterol, LDL, HDL and triglycerides). Assessment items of hematology tests include RBC count, WBC with differential counts, hemoglobin, hematocrit and platelet count. Assessment items of urinalysis include pH, colour, appearance, gravity, erythrocyte, leukocyte, glucose, protein, ketones and nitrite.

   For the ECG test, QTcF must be ≤450msec for females or males, and PR interval <120msec and no evidence of bundle branch block.
7. Willingness of men and women of reproductive potential to observe conventional and highly effective birth control from the beginning of the study screening until 6 months after receiving the last treatment of investigational product. A highly effective method of contraception is defined as follows:

   Highly Effective Methods That Have Low User Dependency
   * Implantable progestogen-only hormone contraception associated with inhibition of ovulation.
   * Intrauterine device (IUD).
   * Intrauterine hormone-releasing system (IUS).
   * Bilateral tubal occlusion.
   * Vasectomized partner (is a highly effective contraceptive method provided that the partner is the sole sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used. The spermatogenesis cycle is approximately 90 days.

   Highly Effective Methods That Are User Dependent (must be used in combination with a male or female condom)
   * Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal, injectable.
   * Progestogen-only hormone contraception associated with inhibition of ovulation: oral, injectable.
8. WOCBP must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study.
9. Males must not donate sperm for at least 90 days after the last dose of study drug.
10. Participants are a current non-smoker (and has not smoked in the 6 months prior to baseline) and will not smoke throughout the course of the study. Screening cotinine test must be negative.

    Additional Inclusion criteria for Phase Ib (Study 2-1, AD participants):
11. Participants who are diagnosed with mild to moderate atopic dermatitis for ≥3 months prior to screening based on the Hanifin and Rajka Criteria. Mild to moderate AD is defined as BSA 2-20%; EASI 3-16; IGA 2 - 3 at both the screening and Day 1 visit.
12. Participants with a Target Area of Atopic Dermatitis of approx. 10 x 10cm on any part of the body other than the scalp, face, palms of hands, soles of feet, buttocks or groin to apply the Study Drug. The Target Lesion Area score needs to be between mild (2) to moderate (3) on the Disease Affected Eczema Area and Severity Indices (EASI) at screening and Day 1.
13. Participant is able to apply the study drug to the Target Lesion Area; or if the Target Lesion is not easily reached (i.e. on their back), has someone who is willing and able to apply the study drug as prescribed during the treatment period.
14. Participants who agree to discontinue all treatment used for their AD, such as topical antihistamines, topical antimicrobials, topical or oral corticosteroid, systemic immune modulating agents and light treatments, as well as bleach baths and avoid prolonged sun exposure during the study period for/on the affected site(s) (except the standard medication oral antihistamine levocetirizine and rescue medication prescribed by the study Investigator(s)). Participants who are taking oral antihistamines need to be on a stable dose for at least 2 months.
15. Participants are required to stop using prohibited topical treatments for at least 14 days before the first investigational drug dose administration (or longer if the treatment half-life requires so 5 half-lives should have elapsed) and prohibited systemic treatment drugs for 28 days before the first investigational drug dose administration (or longer if the treatment half-life requires so 5 half-lives should have elapsed).

    Additional Inclusion criteria for Phase Ib (Study 2-2, RA participants):
16. Diagnosed with Rheumatoid arthritis (RA) prior to screening who fulfil the 2010 ACR/EULAR classification for RA.
17. Mild to moderate disease activity at screening (DAS 28-CRP ≤ 4.5 and ≥ 2.6).
18. Active RA in one Target Joint of either hand or wrist at screening and baseline where both swelling and tenderness/pain is present.

Exclusion Criteria:

Phase Ia and Ib:

1. Participants with conditions at the study drug application site(s) that would interfere with the study drug administration, skin assessment, or reaction to study drug.

   For example: presence of open sores; obvious differences in skin color between applications sites/discolouration such as vitiligo; excessive hair; scar tissue; tattoo.
2. Participants with any unstable health status, defined as having newly diagnosed medical conditions or symptoms of a medical condition that is not yet diagnosed within 30 days prior to the first dose of the study drug.
3. Healthy participants and RA participants only (i.e. does not apply to AD participants): Participants with any diagnosed dermatological condition within 180 days prior to the first study dose.
4. History of anaphylaxis.
5. Participants with any clinically significant (as judged by the Investigator) hematological, endocrine, cardiovascular, hepatic, renal, gastrointestinal, and/or pulmonary disorder.
6. Uncontrolled disease states, such as asthma, psoriasis or inflammatory bowel disease where flares are commonly treated with oral or parenteral corticosteroids.
7. Participants with any predisposing condition that might interfere with the absorption, distribution, metabolism and excretion of the study medication.

   This includes a screening eGFR <60mL/min/1.73m2 or screening transaminases > 1.5 x ULN.
8. Participant had participated in any investigational drug trial and took any investigational drug within 60 days prior to the first study dose.
9. Participant had blood donation of more than 250 mL within 60 days or 500 mL within 90 days prior to the first study drug dose.
10. Participant has current drug abuse or alcohol abuse per Investigator judgement. Participants must have a negative drug and alcohol test at screening and day 1.
11. Participants who are inappropriate to participate in this study, as judged by the Investigator.
12. Participants with any history of or current unstable mental health condition or any lifetime history of suicidal behaviour, as per Investigator judgement.
13. Participants who have known hypersensitivity to the study medication.
14. Participants who are pregnant or breast-feeding or intend to become pregnant during the course of the treatment and follow-up periods.
15. Any history of malignancy of any organ system (other than cervical carcinoma in situ or non-melanoma skin cancers that have been excised) within 5 years prior to study entry.
16. Major surgery (including joint surgery) within 8 weeks prior to screening or during the course of the study.
17. Known active current, or recent history within 3 months, requiring treatment of bacterial, viral, fungal, mycobacterial or other infections.
18. Vaccinated or exposed to a live or attenuated vaccine within the 6 weeks prior to the first dose of study drug, or is expected to be vaccinated or to have household exposure to these vaccines during treatment or up until the follow-up visit.
19. A history (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
20. Any history of any blood clots or clotting disorders (e.g. Deep Vein Thrombosis, Pulmonary Embolism, coagulopathy).
21. Any known immunodeficiency disorder.
22. Mycobacterium tuberculosis (TB) infection as follows:

    * A positive QuantiFERON TB test within the 12 weeks prior to screening or during screening.
    * Any chest imaging (e.g. x-ray, CT) taken at screening or within the 12 weeks prior to screening with changes suggestive of active TB.
    * Been treated or is currently being treated for active or latent TB infection.
    * A history of either untreated or inadequately treated latent or active TB infection.

    Participants with an indeterminate QuantiFERON TB test can have the test repeated and if a negative result is obtained, enrollment may proceed. If the repeat is indeterminate again, the participant will be excluded.
23. Participants who have been tested positive for the following tests:

    * Human immunodeficiency virus (HIV)
    * Hepatitis B virus (HBV): HBsAg or anti-HBc
    * Hepatitis C virus (HCV)

    Additional exclusion criteria for Phase Ib (Study 2-1, AD participants):
24. Participants with active forms of dermatological conditions such as contact dermatitis, seborrheic, discoid, gravitational, asteatotic and dyshidrotic eczema) or other inflammatory skin diseases that are not AD, such as psoriasis, viral infection, fungal infection or bacterial infection.
25. Participants who are inevitable to engage in activities involving excessive or prolonged exposure to sunlight.
26. Treatment with a biologic agent or JAK inhibitor at any time prior to baseline.

    Additional exclusion criteria Phase Ib (Study 2-2, RA participants):
27. Rheumatic autoimmune disease other than rheumatoid arthritis.
28. Functional class IV American College of Rheumatology (ACR) Classification.
29. Prior history of or current inflammatory joint disease other than rheumatoid arthritis (including but not limited to gout, systemic lupus erythematosus, psoriatic arthritis, axial spondylarthritis, reactive arthritis, overlap connective tissue disease). History of secondary Sjogren's syndrome is permitted.
30. Treatment with a biologic agent or JAK inhibitor at any time prior to baseline.

    Note:

    Treatment with traditional DMARDs is allowed provided that the dose is stable for ≥3 months prior to baseline.

    Oral corticosteroids (e.g. Prednisolone) are allowed if the dose is ≤10mg per day and has been stable for two weeks prior to baseline.

    NSAIDs and other low-potency analgesics are allowed if the dose has been stable for two weeks prior to baseline. High potency analgesics are excluded.
31. Intraarticular or parenteral corticosteroids within 6 weeks prior to baseline.
32. Previous treatment with tocilizumab.
33. History of or currently active primary or secondary immunodeficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence and severity of Treatment-Emergent Adverse Events [Safety and Tolerability]. | 1 year
  Assess incidence and severity of treatment-emergent adverse events as determined by CTCAE v5.0 The incidence, nature, and severity of AEs/SAEs including relationship to study treatment from MAD initial study drug administration time of randomisation until Day 14 for MAD participants.
  The incidence, nature, and severity of AEs/SAEs leading to treatment discontinuation from MAD initial study drug administration time of randomisation until Day 7 for MAD participants.
  Clinically significant changes in laboratory parameters, vital signs, 12-lead ECG, and other safety assessments from initial study drug administration time of randomisation until Day 7 for SAD participants.
  Clinically significant changes in laboratory parameters, vital signs, 12-lead ECG, and other safety assessments from MAD initial study drug administration time of randomisation until Day 14 for MAD participants.
To determine the maximum tolerated dose (MTD) of MH004 topical cream. | 1 year
  The determination of the maximum tolerated dose for phase 2.
To establish the recommended phase 2 dose (RP2D). | 1 year
  The determination of RP2D for phase 2 according to the result of dose expansion

SECONDARY OUTCOMES:
Characterization of Pharmacokinetics (Cmax) | Up to 6 Months
  Maximum drug concentration (Cmax)
Characterization of Pharmacokinetics (AUC) | Up to 6 Months
  Area Under the Curve (AUC)
Characterization of Pharmacokinetics (CL) | Up to 6 Months
  Clearance (CL)
Characterization of Pharmacokinetics (t1/2) | Up to 6 Months
  Elimination half-life (t1/2)
Change from baseline Target Lesion EASI score | 1 year
  Percentage of Participants Achieving EASI50，EASI75，EASI90 from Baseline. The EASI50 is defined as a ≥ 50% improvement from baseline in EASI score. The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score. The EASI90 is defined as a ≥ 90% improvement from baseline in the EASI score.
Change from baseline Target Joint swelling and tenderness score | 1 year
  Change from baseline Target Joint swelling and tenderness score by visual anabg scale（VAS）on Day7, Day14 and Day 28 in participants with mild to moderaterheumatoid arthritis.The VAS score runs from 0 to 10, with higher scores indicating worse outcome